CLINICAL TRIAL: NCT03369522
Title: Development of an Epileptic Seizure Detection Algorithm by Continuous Analysis of the Electrocardiogram
Acronym: EPICARD
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_69; 2017-A00114-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2020-09

CONDITIONS: Seizures; Epilepsy; Electrocardiography
Keywords: seizure detection
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Construction: 100 recordings that will be used for the algorithm development
- Validation: 100 recordings for the validation of the algorithm

SUMMARY:
The aim of our project is to develop an epileptic seizure detection algorithm based on the the continuous analysis of the Electrocardiogram

DETAILED DESCRIPTION:
In a first step, the team will build a multi-parametric algorithm on existing records issued from the Epilepsy Monitoring Units. Each selected record will be analyzed by EMU medical team in order to detect seizure on the EEG. The algorithm will adapt in order to obtain the best sensitivity and specificity regarding seizure detection.

in a second step,algorithm will validate on a cohort of other recordings in patients with epilepsy

ELIGIBILITY:
Inclusion Criteria:

* patients with epilepsy
* with a long-term video-EEG recording
* 1 (or more) seizure (s) recorded
* onset seizure clearly defined on the basis of the EEG

Exclusion Criteria:

* bad quality of the Electrocardiogram recording
* pace-maker
* non sinus rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with epilepsy for whom a long-term video-EEG monitoring is required as part of their management
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
ROC curve for seizure detection | 24 months
  ROC curve gives the relation between detection probability and false alarm probability of the algorithm that will be developped

SECONDARY OUTCOMES:
Time of detection of seizures | 24 months
  Time of detection of seizures by the algorithm
ROC curve for Psychogenic seizure detection | 24 months
  ROC curve for Psychogenic seizure detection

CONTACTS AND LOCATIONS:
Overall Officials: William Szurhaj, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - Ch Bethune, Béthune
  - Hôpital Roger Salengro, CHU, Lille
  - Chu Amiens Salouël, Salouël
  - Ch de Valencienne, Valenciennes